CLINICAL TRIAL: NCT00645073
Title: A Phase IV Comparative Study of the Safety and Efficacy of Cefdinir and Levofloxacin for the Treatment of Subjects With Acute Bacterial Sinusitis
Brief Title: Study of the Safety and Efficacy of Cefdinir and Levofloxacin for the Treatment of Subjects With Acute Bacterial Sinusitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Angela M Nilius, PhD, Abbott
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M03-628
Record Dates: First submitted 2008-03-22; First posted 2008-03-27 (Estimated); Last update posted 2008-03-27 (Estimated); Status verified 2008-03

CONDITIONS: Acute Bacterial Sinusitis
Keywords: Acute Bacterial Sinusitis
MeSH Terms: interventions — Cefdinir; Levofloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- A (Active Comparator)
  Interventions: Drug: cefdinir (Omnicef)
- B (Active Comparator)
  Interventions: Drug: levofloxacin

INTERVENTIONS:
Drug: cefdinir (Omnicef) — Two 300 mg cefdinir capsules on Study Days 1-10.
  Other Names: ABT-198; Omnicef; cefdinir
  Arms: A
Drug: levofloxacin — Two 250 mg levofloxacin capsules on Study Days 1-10
  Arms: B

SUMMARY:
To compare the safety and efficacy of a ten-day course of therapy of cefdinir, 600 mg QD, to a ten-day course of therapy of levofloxacin, 500 mg QD, in the treatment of acute bacterial sinusitis.

ELIGIBILITY:
Inclusion Criteria:

* A female must be non-lactating, non-breastfeeding and at no risk for pregnancy.
* A condition of general good health, based upon the results of a medical history, physical examination, and laboratory profile.
* Subject must have a diagnosis of acute bacterial sinusitis. The diagnosis must be based on the following:

  * a sinus radiograph or CT scan performed within 48 hours pre-treatment
  * with evidence of maxillary opacification or air/fluid levels
* Purulent discharge from the nose
* At least one of the following clinical signs and symptoms of acute bacterial sinusitis

  * Lasting for more than 7 days prior to and no longer than 21 days before Evaluation 1: facial pain over the sinus or facial pressure over the sinus or facial tightness over the sinus or facial swelling or toothache.
* Subject must be a suitable candidate for oral antimicrobial therapy and is able to swallow capsules intact.

Exclusion Criteria:

* Subjects who have: chronic sinusitis (signs and symptoms lasting greater than 28 days prior to Evaluation 1)
* Significant anatomical abnormalities of the sinuses
* Any other infection or condition which necessitates use of a concomitant systemic antimicrobial.
* History of any hypersensitivity or allergic reactions to penicillins, cephalosporins (including cefdinir), or quinolones (including levofloxacin).
* Subject who has taken: a systemic antibiotic within 14 days before study drug administration; a long acting injectable antibiotic (e.g., penicillin G benzathine) within 30 days before study drug administration.
* Known significant renal or hepatic impairment.
* Evidence of uncontrolled clinically significant cardiovascular, pulmonary, metabolic, gastrointestinal, neurological or endocrine disease, malignancy, or other abnormality (other than the disease being studied).
* Investigator considers the subject unsuitable for cefdinir or levofloxacin therapy, for any reason.
* Previous enrollment in this study.
* Any underlying condition or disease state that would interfere with the completion of the study procedures and evaluations or absorption of study drug.
* Subject who is currently receiving or who is likely to require any of the following medications during the period between Evaluation 1 (initial presentation to office/clinic) and Evaluation 3 (or within 48 hours after the last dose of study drug): Concomitant theophylline or any theophylline analog, unless plasma levels of these drugs can be adequately monitored during the study; Warfarin and probenecid.
* Immunocompromised subjects.
* Subject who requires parenteral antibiotic therapy for this infection or who has any other infection or condition, that necessitates use of a concomitant systemic antibiotic.
* Subjects receiving antacids containing magnesium, or aluminum, as well as sucralfate, metal cations such as iron, and multivitamin preparations with zinc within 2 hours before or after dosing with study drug.
* Subjects with a known or suspected central nervous system disorder that may predispose the subject to seizures or lower the seizure threshold.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 271 (Actual)
Dates: Start 2003-11; Primary Completion 2004-03 (Actual)

PRIMARY OUTCOMES:
Clinical cure rate | 26 days

SECONDARY OUTCOMES:
Radiographic response | 26 days
Changes from baseline in clinical signs and symptoms | 26 days

CONTACTS AND LOCATIONS:
Locations (25):
- United States (19):
  - Birmingham, Alabama
  - Columbiana, Alabama
  - Eclectic, Alabama
  - Tuscaloosa, Alabama
  - Mesa, Arizona
  - Fresno, California
  - Murray, Kentucky
  - Portage, Michigan
  - Eugene, Oregon
  - Lake Oswego, Oregon
  - Orangeburg, South Carolina
  - Kingsport, Tennessee
  - Milan, Tennessee
  - Corsicana, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - West Jordan, Utah
  - Winchester, Virginia
  - Spokane, Washington
- Poland (6):
  - Gorzów Wielkopolski
  - Krakow
  - Lodz
  - Przybysławice
  - Skierniewice
  - Szczecin